CLINICAL TRIAL: NCT04258514
Title: The Effect of Virtual Reality on Anxiety During Vasectomy
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Similar study published prior to beginning enrollment and we did not anticipate adding new information based on that study
Sponsor: University of Nebraska (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 0034-20-EP
Record Dates: First submitted 2020-01-31; First posted 2020-02-06 (Actual); Last update posted 2023-08-15 (Actual); Status verified 2023-08

CONDITIONS: Vasectomy; Virtual Reality

STUDY DESIGN:
Masking Description: cannot make due to either wearing or not wearing the VR device
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Virtual Reality Vasectomy (Experimental): This group of men will undergo vasectomy while wearing VR goggles.
  Interventions: Procedure: Virtual Reality during vasectomy
- Standard Vasectomy (Experimental): This group of men will undergo a standard vasectomy without using VR goggles.
  Interventions: Procedure: Standard Vasectomy

INTERVENTIONS:
Procedure: Virtual Reality during vasectomy — Virtual Reality
  Arms: Virtual Reality Vasectomy
Procedure: Standard Vasectomy — No Virtual Reality
  Arms: Standard Vasectomy

SUMMARY:
The primary purpose of the study is to determine if the use of Virtual Reality (VR) goggles reduces the degree of anxiety patients experience during vasectomy procedures. The eligibility criteria include a.) appropriate age (19-100 years); b.) undergoing elective vasectomy procedure for purpose of desired sterility; c.) acceptance of wearing goggles; d) able to provide informed consent.There will be two groups, Group A will wear VR goggles and Group B will not. Evaluations will be done by survey to include questions regarding the level of anxiety experienced during the procedure, along with satisfaction scores of the experience.

DETAILED DESCRIPTION:
1. The aim of the study is to evaluate the efficacy of virtual reality goggles (VRG) for improving the patient's experience during vasectomy procedure.
2. The secondary aim is to determine if VRG reduces the level of anxiety experienced during vasectomy procedure.

VR is an immersive, multisensory experience in a three-dimensional environment designed to replicate a real world. It has been shown in multiple studies to decrease acute and chronic pain in a variety of clinical settings. The mechanism is due to distraction by activating visual, auditory and proprioceptive senses. One example of this is a report by G. Pooja et. al. where in VR goggles reduced pain and medication use during orthopedic procedures (1). Another study found decrease in pain in medically treated patients (n=50 patients in 2 groups) after a 15 minute VR viewing on pain reduction compared to 2 -D viewing (2).

ELIGIBILITY:
Inclusion Criteria:

1. Appropriate age range (19-100 years)
2. Undergoing elective vasectomy procedure in the urology clinic
3. Willing to sign consent to participate in the study

Exclusion Criteria:

1. Visually impaired (blind)
2. 18 years of age or younger
3. Subjects under the influence of medications will not be approached regarding study participation.

Ages: 19 Years to 100 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes — only men have vasectomy.
Enrollment: 0 (Actual)
Dates: Start 2021-04-01 (Actual); Primary Completion 2021-06-23 (Actual); Study Completion 2021-06-23 (Actual)

PRIMARY OUTCOMES:
Procedure anxiety | during vasectomy Procedure
  Procedure anxiety measured by Beck Anxiety Inventory
Procedure anxiety | 10 minutes prior to procedure start
  Procedure anxiety measured by Beck Anxiety Inventory
Procedure anxiety | 10 minutes after procedure ends
  Procedure anxiety measured by Beck Anxiety Inventory

CONTACTS AND LOCATIONS:
Overall Officials: Christopher M Deibert, MD, MPH, Principal Investigator — University of Nebraska

IPD SHARING:
Plan to Share IPD: No